CLINICAL TRIAL: NCT01334060
Title: WT1 Immunity Via DNA Fusion Gene Vaccination in Haematological Malignancies by Intramuscular Injection Followed by Intramuscular Electroporation
Acronym: WIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other); Inovio Pharmaceuticals (Industry); Efficacy and Mechanism Evaluation (EME) Programme (Other); Leukemia Research Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHMCAN0700; 2009-017340-14 (EudraCT Number); ISRCTN62678383 (Registry Identifier: NCRN)
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Leukaemia (Acute); Leukaemia (Chronic); Leukaemia (Acute Myeloid); Leukaemia (Acute Lymphoblastic); Leukaemia (Acute Promyelocytic)
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CML HLA A2- (No Intervention)
- AML HLA A2- (No Intervention)
- AML HLA A2+ (Experimental)
  Interventions: Biological: p.DOM-WT1-37 DNA Vaccine and p.DOM-WT1-126 DNA Vaccine
- CML HLA A2+ (Experimental)
  Interventions: Biological: p.DOM-WT1-37 DNA Vaccine and p.DOM-WT1-126 DNA Vaccine

INTERVENTIONS:
Biological: p.DOM-WT1-37 DNA Vaccine and p.DOM-WT1-126 DNA Vaccine — p.DOM-WT1-37: 1mg/dose/vaccine p.DOM-WT1-126: 1mg/dose/vaccine The DNA vaccine will be administered 6 times at 4 weekly intervals. Responders (Immunological but without molecular progression) may continue vaccination 3 monthly to maximum of 24 months. The vaccines will be injected intramuscularly (im) followed by electroporation (EP) into separate locations.
  Arms: AML HLA A2+; CML HLA A2+

SUMMARY:
The study is not currently recruiting new subjects due to an interruption in funding from its sponsors. Efforts are under way to re-establish funding, however, the study is currently on-hold pending the outcome of these re-funding efforts. There have been no safety concerns identified during the study

This is an open label, single dose level, phase II study in two patient groups (CML and AML) using genetic randomisation. Consented and eligible HLA A2+ve patients will be vaccinated with two DNA vaccines and HLA A2 -ve patients will be followed up with molecular monitoring only. The objectives are to evaluate: 1) Molecular response following p.DOM-epitope DNA vaccination in patients with CML (BCR-ABL, WT1) and AML (WT1) at weeks 4, 8, 12, 16, 20 and at months 6, 12, 18 and 24. 2) Time to disease progression, 2 year survival rate (patients with AML) 3) Correlation of molecular responses with immunological responses. Primary Objective: CML: Molecular response of BCR-ABL. AML: Time to disease progression. Secondary Objective: Molecular response of WT1 transcript levels, immune responses to WT1 and DOM, Toxicity, CML-Time to disease progression, next treatment and survival, AML-2 year survival, overall survival

ELIGIBILITY:
Inclusion Criteria:

* CML patients:

Philadelphia chromosome positive CML in chronic phase, in complete cytogenetic response (CCyR) but with detectable BCR-ABL transcripts and maintained the CCyR on imatinib monotherapy for a minimum of 24 months

AML patients:

WT1+ AML in CR or morphologic CR with incomplete blood count recovery (CRi);

All patients:

* ≥ 18 years of age, written informed consent
* Performance status of 0 or 1.
* for vaccination groups: HLA-A0201 positive in at least one allele
* for control groups: HLA A2 negative in both alleles
* renal function and liver function (Creatinine <1.5 x upper limit of normal, liver function tests < 1.5 x upper limit of normal); Lymphocyte count > 1.0 x109/l; normal clotting
* HB>100 g/l
* Adequate venous access for repeated blood sampling according to protocol schedule.
* If sexually active and possibly fertile, patients must agree to use appropriate contraceptive methods during the trial and for six months afterwards.

Exclusion Criteria:

* CML patients:

  * CML in accelerated phase or blast crisis or having achieved CMR at any point during imatinib therapy.
  * Imatinib dose modification in the previous year, Imatinib interruption for more than 15 days in the previous 6 months to enrolment
  * Prior interferon-α therapy
  * hypocellular bone marrow (<20%)
  * Complete molecular response (CMR)

AML patients:

* AML in haematological relapse or eligible for allogeneic SCT.
* hypocellular bone marrow (<20%)
* AML patients with the "good-risk" abnormalities comprised by the core binding factor leukaemias (i.e., AML with the translocation (8;21) and inversion of chromosome 16, and acute promyelocytic leukaemia with the translocation (15;17))

All patients:

* Systemic steroids or other drugs with a likely effect on immune competence are forbidden during the trial. The predictable need of their use will preclude the patient from trial entry
* Major surgery in the preceding three to four weeks from which the patient has not yet recovered.
* Patients who are of high medical risk because of non-malignant systemic disease, as well as those with active uncontrolled infection.
* Patients with any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial, such as concurrent congestive heart failure or prior history of New York Heart Association (NYHA) class III/ IV cardiac disease
* Current malignancies at other sites, with the exception of adequately treated basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for five years and are deemed at low risk for recurrence, are eligible for the study.
* Patients who are serologically positive for or are known to suffer from Hepatitis B, C, Syphilis or HIV. Counselling will be offered to all patients prior to testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02-26 (Actual)

PRIMARY OUTCOMES:
Molecular response following p.DOM-epitope DNA vaccination in patients with CML (BCR-ABL, WT1) and AML (WT1) | 2 years

SECONDARY OUTCOMES:
CML-Time to disease progression, next treatment and survival | 2 years
AML-2 year survival, overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Imperial College NHS Trust, London
  - Southampton University Hospitals NHS Trust, Southampton

REFERENCES:
- [Result] Chaise C, Buchan SL, Rice J, Marquet J, Rouard H, Kuentz M, Vittes GE, Molinier-Frenkel V, Farcet JP, Stauss HJ, Delfau-Larue MH, Stevenson FK. DNA vaccination induces WT1-specific T-cell responses with potential clinical relevance. Blood. 2008 Oct 1;112(7):2956-64. doi: 10.1182/blood-2008-02-137695. Epub 2008 May 23. PMID 18502835
- [Result] Rice J, Ottensmeier CH, Stevenson FK. DNA vaccines: precision tools for activating effective immunity against cancer. Nat Rev Cancer. 2008 Feb;8(2):108-20. doi: 10.1038/nrc2326. PMID 18219306